CLINICAL TRIAL: NCT01251393
Title: Cocaine/Crack Dependence: A Study of the Possible Reduction of Compulsion Under the Use of Biperiden
Brief Title: Cocaine/Crack and Reduction of Compulsion With Biperiden
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Nacional Conseling of Scientific Development and Technology (Other)
Responsible Party: Principal Investigator, Jose Carlos Fernandes Galduroz MD, Dr., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACJC2010
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Cocaine Dependence
Keywords: Cocaine; crack; treatment; dependence; biperiden
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Biperiden; Psychotherapy, Group

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biperiden (Experimental): Thirty volunteers will take three pills of Biperiden (6mg/day) during two months.
  Interventions: Drug: Biperiden
- Placebo (Placebo Comparator): Thirty volunteers will take three pills of Placebo (6mg/day) during two months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Biperiden — Thirty volunteers will take three pills of Biperiden (6mg/day) during two months.
  Other Names: Group psychotherapy
  Arms: Biperiden
Drug: Placebo — Thirty volunteers will take three pills of Placebo (6mg/day) during two months.
  Other Names: Group psychotherapy
  Arms: Placebo

SUMMARY:
Considering the effects of the cholinergic system on the drug reward and self-administration mechanisms, acetylcholine (Ach) may play an important role on cocaine dependence process. Then the present study aims to evaluate biperiden efficacy (a cholinergic antagonist) in attenuate compulsion, one o the main symptoms of the drug dependence.

DETAILED DESCRIPTION:
Cocaine consumption affects around 13.4 mi people or 0.3% of the world population between 15 and 64 years old. The drug dependence has been described by many authors as a dysfunction of the brain reward system. Considering the effects of the cholinergic system on the drug reward and self-administration mechanisms, acetylcholine (Ach) may play an important role on cocaine dependence process. Then the present study aims to evaluate biperiden efficacy (a cholinergic antagonist) in attenuate compulsion, one o the main symptoms of the drug dependence. To accomplish this purpose 60 cocaine or crack male users between 18 and 50 years old will be study. This is a double-blind controlled and randomized placebo study. All the patients will be treated with brief intervention therapy (BIT), and half of them will receive biperiden (6mg/day) while the other half will receive placebo. The treatment efficacy will be evaluated through the comparison between the values obtained on the following measures before and after the treatment: Craving scale of Minnesota and Cocaine/crack consumption questionnaire, and the presence of the cocaine metabolite (benzoylecgonine) on urine.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine or crack dependence, according to the DSM-IV criteria (APA, 1994)

Exclusion Criteria:

* Being under treatment with psychoactive drugs
* Have been diagnosed for other Psychiatric Disorders
* Have dependence diagnosis for other drugs, except for tabacco

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José C F. Galduróz, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- UDED - Drug Dependence Unit, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 participants in the placebo group and 56 participants in the biperiden group.
Period: Overall Study
Arm/Group | Biperiden | Placebo
Started | 56 | 55
Completed | 24 | 11
Not Completed | 32 | 44

BASELINE CHARACTERISTICS:
Groups:
- Biperiden: 55 participants took biperidene for 2 months.
- Placebo: 55 participants took placebo for 2 months.
- Total: Total of all reporting groups
Arm/Group | Biperiden | Placebo | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (7.6) | 31.5 (6.6) | 32.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 56 | 55 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 55 | 111
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 56 | 55 | 111

OUTCOME MEASURES:

1. Primary Outcome: Compulsion
Description: The patients answered the Minnesota Cocaine Craving Scale (Halikas et al., 1991).
  INTENSITY: Evaluation of crack strength by cocaine in the previous week:
  Zero (no craving)---------------------------- -----10 (Intense craving)
  Ranges from 0 to 10 (zero = no craving; 10 intense craving). Using a rule starting from 0, we determine the number that corresponds to the compulsion. The farther from 0 the more intense the compulsion will be.
  Frequency of craving onset: How many times a day 0 time/day - check: 0 point
  1. time/day - check: 1 point
  2. times/day - check: 2 points
  3. to 5 times/day - check: 3 points
  6 to 10 times/day - check: 4 points 11 to 20 times/day - check: 5 points more than 20 times/day - check: 6 points
  Ranges from 0 to 6 points (zero = no craving; 1-2 points: Light; 3-4 points: moderate; 5- 6: intense craving).
  The sum of the points of the subscales provides the final score.
Time Frame: 3 months
Population: A total sample of 166 patients was evaluated during the project. Of that number, 55 did not fulfil the inclusion criteria. The main reasons for exclusion were the presence of clinical comorbidities (active hepatitis, tuberculosis under treatment and epilepsy) or psychiatric comorbidities.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biperiden | Placebo
Number analyzed (Participants) | 56 | 55
score on a scale | 5.9 (2.6) | 5.5 (2.6)
Statistical Analysis 1: Comparison: Biperiden vs Placebo; We evaluated the normality (Kolmogorov's test) and homogeneity (Levene's test) of the sample; Test type: Equivalence — The comparisons between the placebo and the biperiden groups at baseline were performed by means of the independent t-Test. We evaluated the normality (Kolmogorov's test) and homogeneity (Levene's test) of the sample. We used an ANOVA for repeated measures, followed by Bonferroni's post-hoc test to evaluate the efficacy of biperiden in reducing consumption of cocaine/crack; p < 0.05, ANOVA — We used an ANOVA for repeated measures, followed by Bonferroni's post-hoc test to evaluate the efficacy of biperiden in reducing consumption of cocaine/crack

ADVERSE EVENTS:
Groups:
- Placebo; Biperiden: No adverse event
Arm/Group | Placebo | Biperiden
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Biperiden (N=56)
(Nervous system disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes